CLINICAL TRIAL: NCT00399022
Title: Treatment With Duloxetine for OCD Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding was not recieved
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Prof. Joseph Zohar, Chaim Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHEBA-06-4360-JZ-CTIL
Record Dates: First submitted 2006-11-13; First posted 2006-11-14 (Estimated); Last update posted 2008-01-31 (Estimated); Status verified 2008-01

CONDITIONS: OCD
MeSH Terms: interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Outcomes Assessor

INTERVENTIONS:
Drug: Duloxetine

SUMMARY:
Testing the efficacy of the SNRI medication Duloxetine for treating OCD patients who did not respond to SSRI

ELIGIBILITY:
Inclusion Criteria:

* OCD as main diagnosis according to DSM-IV
* Age 18 to 65
* Men and women
* YBOCS score is 18 or more, or 12 or more in case of only obsessions

Exclusion Criteria:

* Patients treated with Duloxetine, currently or in the past
* Patients having comorbid schizophrenia or psychotic disorder or bipolar disorder Patients with substance abuse disorder in the last 6 months Patients who were suicidal or did serious suicide attempt in the last year Pregnant or lactating women, or woman of childbearing potential, which is not using adequate contraception Patients with neurologic disturbance or disorder Patients with serious or imbalanced medical condition Patients with allergic response to SSRI or duloxetine Patients who started new treatment (CBT or pharmacology) in less than 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Zohar, MD, Principal Investigator — Chaim Sheba Medical Center
Locations (1):
- Chaim Sheba Medical Center, Ramat Gan, Israel